CLINICAL TRIAL: NCT04372277
Title: Open Label Study, Evaluating Taltz in Combination With Enstilar (Calcipotriene and Betamethasone Dipropionate) Foam in Psoriasis Patients
Brief Title: Taltz in Combination With Enstilar for Psoriasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC06
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Intervention Model Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Enstilar (Experimental): Enstilar foam
  Interventions: Drug: Enstilar

INTERVENTIONS:
Drug: Enstilar — topical Enstilar foam

SUMMARY:
Enstilar in combination with Taltz for plaque psoriasis.

DETAILED DESCRIPTION:
A single center study of 25 subjects to assess the addition of Enstilar Foam in patients receiving Taltz for ≥ 24 weeks with BSA between 3% and 8%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult ≥ 18 years of age;
* Diagnosis of chronic plaque-type
* Body Surface Area between 3%-8%.
* Patient has been treated with Taltz for a minimum of 24 weeks
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options: hormonal contraception; intrauterine device (IUD); tubal ligation; or partner's vasectomy; Male or female condom diaphragm with spermicide, cervical cap with spermicide, or contraceptive sponge with spermicide.
* Subject must be in general good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination
* Able and willing to give written informed consent prior to performance of any study-related procedures.

Exclusion Criteria

-˂3% or >8% BSA

* Patient not receiving Taltz, or receiving Taltz <24 weeks
* Any condition, which would place the subject at unacceptable risk if he/she were to participate in the study.
* Pregnant or breast feeding, or considering becoming pregnant during the study.
* Use of any investigational drug within 4 weeks prior to randomization, or within 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
* Use of oral systemic medications for the treatment of psoriasis within 4 weeks.
* Patient used other topical therapies to treat within 2 weeks of the Baseline Visit.
* Patient received UVB phototherapy within 2 weeks of Baseline.
* Patient received PUVA phototherapy within 4 weeks of Baseline.
* Patient has a known hypersensitivity to the excipients of Enstilar® as stated in the label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Body Surface Area 0 or 1 | 4 weeks
  Body surface area where 1 palm is equivalent to 1%. Endpoint will evaluate number of patiens who achieve body surface are 0 or 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States